CLINICAL TRIAL: NCT01823263
Title: Metabolic and Cognitive Effects of Sleep Deprivation
Brief Title: Metabolic and Cognitive Parameters Following Partial Sleep Deprivation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SleepPartialJCCB2013
Record Dates: First submitted 2013-02-21; First posted 2013-04-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Sleep Deprivation; Sleep
MeSH Terms: conditions — Sleep Deprivation | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partial sleep deprivation (Experimental): Partial sleep deprivation: participants will have a 4-h sleep opportunity before a 'Blood Sample' will be taken, and the 'Memory tasks', 'Working memory function task' and 'Portion size task' will be performed. This will be followed by an 'Interference task', followed by repeated blood sampling and an 'Intake task'.
  Interventions: Behavioral: Portion Size Task; Procedure: Blood sample; Procedure: Interference task; Behavioral: Memory tasks; Behavioral: Intake task; Behavioral: Working memory function task
- Normal sleep (Experimental): Normal sleep: participants will have an 8-h sleep opportunity before a 'Blood Sample' will be taken, and the 'Memory tasks', 'Working memory function task' and 'Portion size task' will be performed. This will be followed by an 'Interference task', followed with repeated blood sampling and an 'Intake task'.
  Interventions: Behavioral: Portion Size Task; Procedure: Blood sample; Procedure: Interference task; Behavioral: Memory tasks; Behavioral: Intake task; Behavioral: Working memory function task

INTERVENTIONS:
Behavioral: Portion Size Task — Participants are given a computer program that gives them the opportunity to choose the portions of a variety of food items that they would ideally like to consume
Procedure: Blood sample — In the morning following partial sleep deprivation or normal sleep, a blood sample will be taken to assess the level of metabolism-linked and neurodegenerative-linked molecules, as well as to assay blood serum and plasma for the presence of hormones involved in hunger such as ghrelin
Procedure: Interference task — 30-minute interference task
Behavioral: Memory tasks — Participants will be allowed to learn a procedural memory task before going to bed. Participants will be retested in the morning to assess their change in performance. Other memory tests will also be given to assess the working memory performance in the morning following the intervention.
Behavioral: Intake task — After a normal night of sleep or partial sleep deprivation, participants are presented with an ad libitum meal choice and can select the amount to ingest during a limited time window. Amount and selection will be recorded
Behavioral: Working memory function task — Participants will be evaluated on their working memory performance in the morning following either nighttime intervention (NS or PSD)

SUMMARY:
The purpose of this study is to determine whether partial sleep deprivation, as compared with normal sleep, influences certain metabolic and cognitive parameters, related to food intake, hunger and memory functions, when participants are shielded from external time cues.

DETAILED DESCRIPTION:
It is predicted that partial sleep deprivation negatively affects the hormonal status, e.g. upregulating ghrelin and other hunger-promoting hunger hormones, while showing impaired memory functions. It is also predicted that participants will tend to increase their desired portion sizes after partial sleep deprivation, compared with after a normal night's sleep.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 20-28y
* Healthy (self-reported) and not on medication
* Non-smoking
* Normal sleep-wake rhythm (i.e. 7-8 h per night, self-reported and verified by sleep diaries)
* Normal dietary habits (regular meal pattern with daily breakfast)

Exclusion Criteria:

* Major illness
* Taking any serious medications
* Any sleep conditions (e.g. irregular bedtimes, sleep complaints)
* Any dietary issues with the food items provided
* A history of endocrine, neurological or psychiatric disorders
* Shift work in the previous 3 months
* Travel over several time zones within the previous two months

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Memory tasks | Change in memory performance between learning (at 2230 hours in NS and PSD condition) before going to sleep, and at 0800 and 0930 hours (following PSD or NS)
  Procedural memory performance after learning a procedural memory task close to going to bed, followed by either partial sleep deprivation (PSD) or normal sleep (NS), and comparing the performance the following morning at two time points. Participants spatial memory performance in the morning at two time points, following PSD will also be compared with that following NS, after having learned such a memory task in the evening before going to bed.

SECONDARY OUTCOMES:
Circulating hormone levels | Change in circulating hormone levels and other metabolism-linked and neurodegeneration-associated molecules at 0730, 0830, 0910, 0925, 0940, 1010, 1040, 1105, and 1150 hours following the respective nighttime intervention and after the interference task
  Interference task given at 0900 hours
Intake task | Change in intake at around 1200 hours, following the respective nighttime intervention (NS or PSD)
  Participants are presented with an ad libitum meal choice and can select the amount to ingest during a limited time window. Amount and selection will be recorded.
Working memory function task | Change in memory performance at 0800 hours and after the interference task again at 0930 hours (between and following PSD or NS)
  Participants will be evaluated on their working memory performance in the morning following either nighttime intervention (NS or PSD) and before and after an interference task
Portion Size Task | Change in selected portion size from baseline (at 0800 hours following the nighttime intervention), to one hour later, i.e. after an interference task
  Participants will be evaluated on their tendency to choose larger or smaller portions of a variety of meal items on a computer screen. This will be conducted both following partial sleep deprivation and normal sleep, and changes before and after a short interference task will be compared between these two conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benedict, PhD, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Department of Neuroscience, Uppsala University, Uppsala, Uppsala County, Sweden